CLINICAL TRIAL: NCT07366450
Title: Safety and Efficacy of High-Intensity Loading Dose Versus Standard Weekly Dosing of Ergocalciferol (Vitamin D2) for Vitamin D Normalization in Patients With Newly Diagnosed Aggressive Non-Hodgkin Lymphoma: A Randomized, Open-Label, Controlled Trial
Brief Title: High-Dose vs Standard Ergocalciferol for Vitamin D Normalization in Aggressive Non-Hodgkin Lymphoma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Phramongkutklao College of Medicine and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Hemato-002
Record Dates: First submitted 2026-01-05; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Vitamin D 25-Hydroxylase Deficiency; Lymphoma Non-Hodgkin
Keywords: Non-Hodgkin lymphoma; Vitamin D deficiency; Overall survival; Efficacy
MeSH Terms: conditions — Vitamin D Hydroxylation-Deficient Rickets, Type 1B; Lymphoma, Non-Hodgkin; Vitamin D Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-Dose Loading Ergocalciferol (Experimental): Participants receive a high-dose loading regimen of ergocalciferol (vitamin D₂) for rapid normalization of serum vitamin D levels, in combination with standard first-line chemoimmunotherapy for aggressive non-Hodgkin lymphoma.
  Interventions: Drug: High-Dose Loading Ergocalciferol
- Standard Weekly Ergocalciferol (Active Comparator): Participants receive standard weekly dosing of ergocalciferol (vitamin D₂) for vitamin D normalization, in combination with standard first-line chemoimmunotherapy for aggressive non-Hodgkin lymphoma.
  Interventions: Drug: Standard Weekly Ergocalciferol

INTERVENTIONS:
Drug: High-Dose Loading Ergocalciferol — Dose and Schedule:
  * Loading phase: Ergocalciferol 20,000 IU orally once daily (1 capsule per dose), administered 1-2 hours before breakfast, for 7 consecutive days.
  * Intensified phase: Following the loading phase, ergocalciferol 20,000 IU orally three times per week (Monday, Wednesday, and Friday) for a total treatment duration of 6 weeks from the first dose.
  * Maintenance phase: After completion of the initial 6-week treatment period, ergocalciferol 20,000 IU orally once weekly (Monday) until completion of lymphoma treatment.
  * Maximum duration of vitamin D₂ administration: Up to 18 weeks from the first dose of ergocalciferol. Thereafter, vitamin D dosing may be adjusted at the discretion of the treating physician.
  Arms: High-Dose Loading Ergocalciferol
Drug: Standard Weekly Ergocalciferol — Dose and Schedule:
  * Standard phase: Ergocalciferol 20,000 IU orally three times per week (Monday, Wednesday, and Friday), administered as 1 capsule per dose, 1-2 hours before breakfast, for a total duration of 6 weeks from the first dose.
  * Maintenance phase: After completion of the 6-week standard dosing period, ergocalciferol 20,000 IU orally once weekly (Monday) until completion of lymphoma treatment.
  * Maximum duration of vitamin D₂ administration: Up to 18 weeks from the first dose of ergocalciferol. Thereafter, vitamin D dosing may be adjusted at the discretion of the treating physician.
  Arms: Standard Weekly Ergocalciferol

SUMMARY:
The goal of this clinical trial is to evaluate whether a high-intensity loading dose of ergocalciferol (vitamin D2) can normalize blood vitamin D levels more rapidly and safely than standard weekly dosing in patients with newly diagnosed aggressive non-Hodgkin lymphoma. The study will also assess the safety of both dosing strategies.

The main questions it aims to answer are:

* Does a high-intensity loading dose of ergocalciferol lead to faster normalization of serum 25-hydroxyvitamin D levels compared with standard weekly dosing?
* Are there differences in safety and adverse events between the two dosing strategies?

Researchers will compare a high-intensity loading dose regimen of ergocalciferol with a standard weekly dosing regimen to determine differences in vitamin D normalization and safety outcomes.

Participants will:

* Be randomly assigned to receive either a high-intensity loading dose or a standard weekly dose of ergocalciferol (vitamin D2)
* Receive standard first-line immunochemotherapy for aggressive non-Hodgkin lymphoma
* Have blood tests to monitor vitamin D levels, calcium, phosphate, and safety parameters at scheduled visits
* Be followed for treatment response, survival outcomes, and adverse events during and after therapy

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 20 years.
* Newly diagnosed aggressive non-Hodgkin lymphoma, confirmed by histopathological examination according to the WHO Classification of Haematolymphoid Tumours, 5th edition, with an indication for standard first-line chemoimmunotherapy
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-3.
* Serum 25-hydroxyvitamin D level < 30 ng/mL within 14 days prior to randomization.
* Adequate organ function to receive full-dose standard chemotherapy.
* Ability to provide written informed consent.

Exclusion Criteria:

* Mild hypercalcemia (corrected Ca > 10.4 mg/dL)
* Hyperphosphatemia (PO4 > 4.5 mg/dL)
* History of urolithiasis associated with hypercalciuria or a diagnosis of primary hyperparathyroidism.
* Chronic kidney disease stage 4 or higher (estimated glomerular filtration rate [eGFR] < 30 mL/min/1.73 m²).
* Inability to take oral medication, active gastrointestinal bleeding, or malabsorption syndrome.
* Pregnancy or breastfeeding.
* Prior systemic therapy for lymphoma.
* Ongoing tumor lysis syndrome requiring urgent treatment.
* Prior use of vitamin D supplements (ergocalciferol or cholecalciferol).

Withdrawal Criteria:

* Development of mild hypercalcemia.
* Development of mild hypophosphatemia.
* Development of hypervitaminosis D.
* Occurrence of severe adverse events (AEs) or side effects for which the investigator considers discontinuation of the study drug necessary for patient safety.
* Investigator's judgment that continued participation may pose a safety risk, such as the occurrence of serious infection, febrile neutropenia, or organ failure.
* Non-adherence to study medication, defined as cumulative vitamin D₂ intake of less than 80% of the expected cumulative dose at the time of serum vitamin D assessment.
* Participant withdrawal of consent to continue participation in the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants Achieving Vitamin D Normalization by Day 21 | Day 21 (± 3 days) after the first dose of study medication
  Vitamin D normalization is defined as a serum 25-hydroxyvitamin D level ≥ 30 ng/mL. This outcome is assessed as a binary outcome (yes/no).

SECONDARY OUTCOMES:
Event-Free Survival (EFS) | Up to 3 years
  Event-free survival is defined as the time from randomization to the first occurrence of disease progression, relapse after response, initiation of new lymphoma therapy, or death from any cause.
Progression-Free Survival (PFS) | Up to 3 years
  Progression-free survival is defined as the time from randomization to the first documented disease progression according to the Lugano 2014 criteria or death from any cause, whichever occurs first.
Overall Survival (OS) | Up to 3 years
  Overall survival is defined as the time from randomization to death from any cause.
Best Overall Response (BOR) | Through the completion of first-line immunochemotherapy, approximately 24 weeks
  Best overall response is defined as the best response achieved after completion of first-line immunochemotherapy, including complete response (CR) or partial response (PR), as assessed by PET-CT or CT scan according to the Lugano 2014 criteria.
Change in Serum 25-Hydroxyvitamin D Level | Day 21 (± 3 days), Day 42 (± 3 days), Day 63 (± 3 days), and Day 126 (± 3 days) (end of treatment)
  Changes in serum 25-hydroxyvitamin D levels will be compared between study arms and summarized as absolute change and central tendency measures (mean or median).
Incidence of Grade ≥ 3 Infections | From randomization through 30 days after the last dose of study treatment, approximately 22 weeks
  Incidence of infections graded ≥ 3 according to the Common Terminology Criteria for Adverse Events (CTCAE), version 6.0.
Safety and Treatment-Related Toxicity | From randomization through 30 days after the last dose of study treatment, approximately 22 weeks
  Safety and toxicity will be assessed based on the incidence of hypercalcemia, hypophosphatemia, and other adverse events, graded according to CTCAE version 6.0.

CONTACTS AND LOCATIONS:
Overall Officials: Tanapun Thamgrang, Principal Investigator — Division of Hematology, Department of Medicine, Phramongkutklao Hospital
Locations (1):
- Phramonkutklao Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to institutional policy and privacy concerns. Only aggregate data may be shared upon reasonable request.